CLINICAL TRIAL: NCT03513198
Title: Changes in Tumor Vascularity Depicted by Contrast-Enhanced Endoscopic Ultrasonography as a Predictor of Treatment Efficacy in Patients With Locally Advanced and Metastatic Pancreatic Cancer (PEACE)
Brief Title: Perfusion Assessment With Contrast-Enhanced EUS in Locally Advanced and Metastatic Pancreatic Cancer
Acronym: PEACE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Medicine and Pharmacy Craiova (Other)
Collaborators: Copenhagen University Hospital at Herlev (Other); Iuliu Hatieganu University of Medicine and Pharmacy (Other); Central Military Hospital Bucharest (Unknown); Ponderas Regina Maria Hospital Bucharest (Unknown); Caritas-Krankenhaus Bad Mergentheim (Other); Helios Kliniken Meiningen (Unknown); University of Santiago de Compostela (Other); Hospital Märkisch Oderland Wriezen/ Strausberg (Unknown); Institut Paoli-Calmettes (Other); Ospedale San Raffaele (Other); University College London Hospitals (Other); Newcastle-upon-Tyne Hospitals NHS Trust (Other); M.D. Anderson Cancer Center (Other); Shengjing Hospital (Other); Asan Medical Center (Other); Tokyo Medical University (Other); Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PEACE
Record Dates: First submitted 2018-02-13; First posted 2018-05-01 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Pancreas Cancer
Keywords: contrast-enhanced endoscopic ultrasound; endoscopic ultrasound elastography; tumor vascularity; prognostic
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Endosonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-resectable pancreatic cancer: All patients with a suspicion of pancreatic masses will undergo EUS (including EUS-FNA for confirmation of diagnosis). A positive cytological diagnosis will be taken as a final proof of malignancy of the pancreas mass. The diagnoses obtained by EUS-FNA will be further verified during a clinical follow-up of at least 6 months.
  Both pancreatic adenocarcinomas and pancreatic neuroendocrine tumors will be included.
  Endoscopic ultrasound (including fine needle aspiration for confirmation of diagnosis) with sequential contrast-enhanced endoscopic ultrasound and elastography endoscopic ultrasound and contrast-enhanced computed tomography will be performed before and 2 months after the first course of treatment
  Interventions: Diagnostic Test: Endoscopic ultrasound (including fine needle aspiration); Other: Contrast-enhanced endoscopic ultrasound (CE-EUS); Other: Endoscopic ultrasound elastography (EG-EUS); Diagnostic Test: Contrast-enhanced computed tomography (CT)

INTERVENTIONS:
Diagnostic Test: Endoscopic ultrasound (including fine needle aspiration) — EUS will be performed before (including EUS-FNA for confirmation of diagnosis) and 2 months after the first course of treatment.
  * Protocol of EUS with EUS-FNA should include linear EUS instruments with complete examinations of the pancreas.
  * Tumor characteristics (echogenicity, echostructure, size) will be described as well as presence/absence of power Doppler signals.
  * EUS-FNA will be performed in all pancreatic masses with at least four passes.
Other: Contrast-enhanced endoscopic ultrasound (CE-EUS) — CE-EUS will be performed during usual EUS examination before and 2 months after the first course of chemotherapy.
  * The starting point of the timer will be considered the moment of intravenous contrast injection (Sonovue 4.8 mL).
  * The whole movie (T0-T120s) will be recorded in a DICOM format on the embedded HDD of the ultrasound system, for later analysis.
  * All post-processing and computer analysis of digital movies will be performed within the coordinating IT Center using Vue-Box
Other: Endoscopic ultrasound elastography (EG-EUS) — EUS-EG will be performed during usual EUS examinations, before and 2-months after the first course of chemotherapy, with two movies of 10 seconds recorded on the embedded HDD
  * The region of interest for EUS-EG will be preferably larger than the focal mass. If the focal mass is larger than 3 cm, part of the mass will be included in the ROI, as well as the surrounding structures. Very large ROI for the elastography calculations will be avoided
  * The following pre-settings will be used in all centers: elastography color map 1, frame rejection 2, noise rejection 2, persistence 3, dynamic rage 4, smoothing 2, blend 50%.
  * SR and SH will be measured; with three measurements made and recorded on the embedded HDD.
Diagnostic Test: Contrast-enhanced computed tomography (CT) — * Contrast-enhanced computed tomography will be obtained before treatment to assess the local extension of the tumor, and presence of lymph nodes and distant metastases.
  * A template will be used to report the imaging results.
  * The template includes morphologic, arterial, venous, and extrapancreatic evaluations.
  * Contrast-enhanced computed tomography will be performed 2 months after the first course of chemotherapy, using the same template, in order to evaluate the tumor response. Tumor response will be assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST).

SUMMARY:
Patients with non-resectable pancreatic cancer have a poor prognosis.The analysis of prognostic factors before treatment may be helpful in selecting appropriate candidates for chemotherapy and determining treatment strategies.

The aim of the PEACE study is to assess the vascularity of pancreatic malignant tumors using contrast-enhanced endoscopic ultrasonography and to clarify the prognostic value of tumor vascularity in patients with locally advanced and metastatic pancreatic cancer.

DETAILED DESCRIPTION:
Introduction and rationale:

Pancreatic cancer (PC) is one of the most lethal and therapeutically resistant malignancies, with a grim prognosis that is attributed to the late clinical presentation and the relative chemoresistance of the disease.

Even with identical chemotherapy regimens, some patients experience improvements in survival and tumor response, whereas other patients only experience inconvenience and increased toxicity. It has been suggested that the burden of treatment should not be added to the suffering of those with advanced pancreatic cancer. Therefore, understanding prognostic factors before treating patients with antitumoral agents may be helpful in selecting those patients predicted to have an improved survival and tumor response after treatment.

Studies have shown that angiogenesis is an important factor that influences the prognostic of solid tumors, including pancreatic tumors. Contrast-enhanced imaging methods can offer detailed information on tumor vascularity. Contrast-enhanced endoscopic ultrasound (CE-EUS) is a new method which allows detailed characterization of focal pancreatic masses. CE-EUS offers high-resolution images of the pancreas that far surpass those achieved by computed tomography, ultrasound, or magnetic resonance imaging. CE-EUS can detect intratumoral vessels in the pancreatic lesions. One of the fluoro-gas-containing contrast agents used in CE-EUS is Sonovue®, which is isotonic, stable and resistant to pressure, with a viscosity similar to blood. It does not diffuse into the extravascular compartment remaining within the blood vessels until the gas dissolves and is eliminated in the expired air (blood pool contrast agent). The safety profile of SonoVue showed a very low incidence of side effects; it is not nephrotoxic and the incidence of severe hypersensitivity is similar to other magnetic resonance imaging contrast agents. Moreover, Sono-Vue is approved for clinical use in European Union countries.

The hypothesis that tumors with intratumoral vessels are chemosensitive appears to be reasonable because drugs penetrate tumors through vessels. Therefore, it is possible that hypoxic condition in tumor tissue leads to chemoresistance and poor prognosis in patients with pancreatic carcinoma who received systemic chemotherapy. However, whether low vascularized tumors correlate with the chemoresistance and poor prognosis is still unclear. Patients with non-resectable pancreatic cancer have an especially poor prognosis and have many severe symptoms.The analysis of prognostic factors before treatment may be helpful in selecting appropriate candidates for chemotherapy and determining treatment strategies. For example, patients who have a poor prognosis may be treated best with only supportive care because of their short survival. Consequently, the aim of the PEACE study is to assess the vascularity of pancreatic malignant tumors with CE-EUS and to clarify the prognostic value of tumor vascularity in patients with advanced PC.

Moreover, studies have shown that angiotensin inhibition enhances drug delivery and potentiates chemotherapy by decompressing tumor blood vessels. Chauchan et al. demonstrated that the angiotensin inhibitor losartan reduces stromal collagen and hyaluronan production. Consequently, losartan reduces solid stress in tumors resulting in increased vascular perfusion. Through this physical mechanism, it can improve drug and oxygen delivery to tumors, thereby potentiating chemotherapy and reducing hypoxia in breast and pancreatic cancer models. Accordingly, another aim of our study will be to examine the correlation between tumor vascularity and angiotensin inhibitors use in patients using these drugs to control arterial hypertension.

Objectives:

Primary Objective:

• to register time-intensity curve (TIC) analysis-derived parameters, obtained from post-processing of CE-EUS recordings with a commercially available software, before and after chemotherapy and to describe tumor changes in vascularity after treatment.

Secondary Objectives:

* to prospectively determine whether the CE-EUS parameters can be used to predict response to treatment in patients with locally advanced and metastatic pancreatic cancer. Tumor response will be assessed by contrast-enhanced computed tomography, according to the Response Evaluation Criteria in Solid Tumors (RECIST)
* to determine the correlation between CE-EUS parameters before treatment and overall survival and progression-free survival
* to determine the correlation between changes in tumor vascularity and progression-free survival and overall survival
* to assess quantitative elastography parameters during EUS, before and after systemic treatment and determine their correlation with overall survival and progression-free survival
* to examine the correlation between tumor vascularity and angiotensin inhibitors use.

Study design:

This is a prospective, non-randomized, single-arm, observational, multicenter study aiming to assess changes in tumor vascularity using CE-EUS before and after systemic treatment in patients with locally advanced and metastatic pancreatic cancer and to examine the correlation between vascular changes and treatment response, progression-free survival and overall survival.

All patients with a suspicion of pancreatic masses will undergo EUS (including endoscopic ultrasound-fine needle aspiration for confirmation of diagnosis), with sequential elastography EUS (EG-EUS) and CE-EUS. A positive cytological diagnosis will be taken as a final proof of malignancy of the pancreas mass. The diagnoses obtained by EUS-fine needle aspiration will be further verified during a clinical follow-up of at least 6 months. Contrast-enhanced computed tomography (CT) will be performed as pretreatment staging study to assess the diagnosis of pancreatic cancer, local extension of the tumor, and presence of distant and lymph node metastasis.

Patients with a confirmed diagnosis of pancreatic cancer (both adenocarcinomas and neuroendocrine tumors will be included) will undergo systemic treatment. Selection of the specific treatment regimen will be according to individual physicians' choice.

Two months after the first course of systemic chemotherapy, CT and EUS (with sequential EG-EUS and CE-EUS) will be repeated. CT will be performed in order to evaluate the tumor response. Tumor response will be assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST).

CE-EUS will be performed during usual EUS examinations, with the whole movie (T0-T120s) recorded in a DICOM format on the embedded HDD of the ultrasound system, for later analysis. In order to minimize human bias, all post-processing and computer analysis of digital movies will be performed within the coordinating IT Center, with all programmers and statisticians being blinded to the clinical, imaging and pathological data. Off-line analysis of time-intensity curves will be performed using Vue-Box, which yields the following quantitative parameters: Peak Enhancement (PE), Wash-in Area Under the Curve (Wi-AUC), Rise Time (RT), mean Transit Time (mTT), Time To Peak (TTP), Wash-in Rate (WiR) and Wash-in Perfusion Index (WiPI). The software also provides referenced values (expressed in percentages), aligning the set of values for the tumor Region of interest (ROI) to the parenchymal ones.

EUS-EG will also be performed during usual EUS examinations, with two movies of 10 seconds recorded on the embedded Hard Disk Drive (HDD) in order to minimize variability and to increase repeatability of acquisition. Strain Ratio (SR) and SH (Strain Histogram) will be measured; with three measurements made and recorded on the embedded HDD.

The patients will be followed-up for at least six months through clinical examination, biological exams and transabdominal ultrasound, eventually with a repeat spiral CT / EUS after six months.

For each patient, the following information will be recorded and uploaded to http://oncobase.umfcv.ro/ (this website aims to provide hosting and support for multicentric studies; all registered users can access the project and submit the data or upload files through a form defined and controlled by the project's coordinator):

* Age
* Gender
* Primary tumor location (pancreatic head or pancreatic body and tail)
* Primary tumor size
* Tumor status (metastatic or locally advanced)
* Site of metastasis
* Histologic grade
* Serum carcinoembryonic antigen (CEA) level
* Serum carbohydrate antigen 19-9 (CA19-9) level
* Prior biliary drainage (presence or absence).
* Antitumoral agent (chemotherapy regimen).
* Angiotensin inhibitors (drug, dose).
* Parameters of the pancreatic cancer CT reporting template
* EUS, CE-EUS, EG-EUS parameters (echogenicity, echostructure, size, presence/absence of power Doppler signals, Strain Ratio, Strain Histogram, Peak Enhancement (PE), Wash-in Area Under the Curve (Wi-AUC), Rise Time (RT), mean Transit Time (mTT), Time To Peak (TTP), Wash-in Rate (WiR) and Wash-in Perfusion Index (WiPI)).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 90 years old, men or women
* Signed informed consent for CE-EUS, EG-EUS and FNA biopsy
* The diagnosis of pancreatic cancer histologically confirmed by fine needle aspiration (FNA) with EUS
* Both pancreatic adenocarcinoma and pancreatic neuroendocrine tumors will be included
* Unresectable, locally advanced and/or metastatic disease.

Exclusion Criteria:

* Previous chemotherapy or radiotherapy
* Resectable pancreatic tumors

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with a confirmed diagnosis of locally advanced/metastatic pancreatic cancer (both adenocarcinoma and neuroendocrine tumors will be included)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Change of Peak Enhancement (PE) from baseline to 2 months after the first course of treatment | baseline and 2 months after the first course of treatment
  PE represents a TIC analysis-derived parameter, obtained from post-processing of CE-EUS recordings with a commercially available software
Change of Wash-in Area Under the Curve (Wi-AUC) from baseline to 2 months after the first course of treatment | baseline and 2 months after the first course of treatment
  Wi-AUC represents a TIC analysis-derived parameter, obtained from post-processing of CE-EUS recordings with a commercially available software
change of Rise Time (RT) from baseline to 2 months after the first course of treatment | baseline and 2 months after the first course of treatment
  RT represents a TIC analysis-derived parameter, obtained from post-processing of CE-EUS recordings with a commercially available software
change of mean Transit Time (mTT) from baseline to 2 months after the first course of treatment | baseline and 2 months after the first course of treatment
  mTT represents a TIC analysis-derived parameter, obtained from post-processing of CE-EUS recordings with a commercially available software
Change of Time To Peak (TTP) from baseline to 2 months after the first course of treatment | baseline and 2 months after the first course of treatment
  TTP represents a TIC analysis-derived parameter, obtained from post-processing of CE-EUS recordings with a commercially available software
Change of Wash-in Rate (WiR) from baseline to 2 months after the first course of treatment | baseline and 2 months after the first course of treatment
  Wir represents a TIC analysis-derived parameter, obtained from post-processing of CE-EUS recordings with a commercially available software
Change of Wash-in Perfusion Index (WiPI) from baseline to 2 months after the first course of treatment | baseline and 2 months after the first course of treatment
  WiPI represents a TIC analysis-derived parameter, obtained from post-processing of CE-EUS recordings with a commercially available software

SECONDARY OUTCOMES:
Overall survival | 1 year
  The overall survival (OS) will be measured from the first day of chemotherapy to the date of death
Progression-free survival | 1 year
  The progression-free survival (PFS) will be measured from the first day of chemotherapy to the date of progressive disease.
Tumor response to treatment | 2 months after the first course of treatment
  Contrast-enhanced computed tomography will be performed 2 months after the first course of chemotherapy in order to evaluate the tumor response.
  Tumor response will be assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST). According to RECIST guidelines,complete response (CR) is defined as the complete disappearance of the tumor, partial response (PR) as ≥30% decrease in longest diameter (LD), progressive disease (PD) as ≥20% increase in LD, and stable disease (SD) as a decrease or increase less than PR or PD based on anatomic assessment. Patients with CR or PR will be defined as responders, whereas those with PD or SD are defined as non-responders.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Saftoiu, MD PhD FASGE, Principal Investigator — University of Medicine and Pharmacy Craiova

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lowenfels AB, Maisonneuve P. Epidemiology and risk factors for pancreatic cancer. Best Pract Res Clin Gastroenterol. 2006 Apr;20(2):197-209. doi: 10.1016/j.bpg.2005.10.001. PMID 16549324
- [Background] Folkman J. What is the evidence that tumors are angiogenesis dependent? J Natl Cancer Inst. 1990 Jan 3;82(1):4-6. doi: 10.1093/jnci/82.1.4. No abstract available. PMID 1688381
- [Background] Fidler IJ, Ellis LM. The implications of angiogenesis for the biology and therapy of cancer metastasis. Cell. 1994 Oct 21;79(2):185-8. doi: 10.1016/0092-8674(94)90187-2. No abstract available. PMID 7525076
- [Background] Ikeda N, Adachi M, Taki T, Huang C, Hashida H, Takabayashi A, Sho M, Nakajima Y, Kanehiro H, Hisanaga M, Nakano H, Miyake M. Prognostic significance of angiogenesis in human pancreatic cancer. Br J Cancer. 1999 Mar;79(9-10):1553-63. doi: 10.1038/sj.bjc.6690248. PMID 10188906
- [Background] Saftoiu A, Vilmann P, Bhutani MS. The role of contrast-enhanced endoscopic ultrasound in pancreatic adenocarcinoma. Endosc Ultrasound. 2016 Nov-Dec;5(6):368-372. doi: 10.4103/2303-9027.190932. PMID 28000627
- [Background] Yamashita Y, Ueda K, Itonaga M, Yoshida T, Maeda H, Maekita T, Iguchi M, Tamai H, Ichinose M, Kato J. Tumor vessel depiction with contrast-enhanced endoscopic ultrasonography predicts efficacy of chemotherapy in pancreatic cancer. Pancreas. 2013 Aug;42(6):990-5. doi: 10.1097/MPA.0b013e31827fe94c. PMID 23851433
- [Background] Sanchez MV, Varadarajulu S, Napoleon B. EUS contrast agents: what is available, how do they work, and are they effective? Gastrointest Endosc. 2009 Feb;69(2 Suppl):S71-7. doi: 10.1016/j.gie.2008.12.004. No abstract available. PMID 19179175
- [Background] Zhang X, Galardi E, Duquette M, Lawler J, Parangi S. Antiangiogenic treatment with three thrombospondin-1 type 1 repeats versus gemcitabine in an orthotopic human pancreatic cancer model. Clin Cancer Res. 2005 Aug 1;11(15):5622-30. doi: 10.1158/1078-0432.CCR-05-0459. PMID 16061881
- [Background] Chauhan VP, Martin JD, Liu H, Lacorre DA, Jain SR, Kozin SV, Stylianopoulos T, Mousa AS, Han X, Adstamongkonkul P, Popovic Z, Huang P, Bawendi MG, Boucher Y, Jain RK. Angiotensin inhibition enhances drug delivery and potentiates chemotherapy by decompressing tumour blood vessels. Nat Commun. 2013;4:2516. doi: 10.1038/ncomms3516. PMID 24084631
- [Background] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437